CLINICAL TRIAL: NCT03684135
Title: Satisfaction Assessment of Patients With Local Breast Cancer When Using Cosmetics During Chemotherapy and Post-treatment Thermal Cure
Acronym: COSMIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-004938-28
Record Dates: First submitted 2018-07-11; First posted 2018-09-25 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Local Breast Cancer Patients
Keywords: Breast cancer; Cosmetics; Satisfaction; Chemotherapy; Thermal cure
MeSH Terms: conditions — Breast Neoplasms; Personal Satisfaction | interventions — Cosmetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of cosmetics during chemotherapy and thermal cure (Experimental): Use of cosmetics during chemotherapy and post-treatment thermal cure
  Interventions: Other: Cosmetics

INTERVENTIONS:
Other: Cosmetics — "Tendre Caresse au cold cream" body cream from Cosmétosource "Crème de douche" face and body cleanser from Cosmétosource

SUMMARY:
The purpose of this study is to assess the satisfaction, the observance, the intolerance, the qualitative appreciation and the expectations of the patients related to the use of the cosmetic products ("Tendre Caresse au cold cream" body cream and "Crème de douche" face and body cleanser from Cosmétosource) during chemotherapy and post-treatment thermal cure

ELIGIBILITY:
Inclusion Criteria:

* Woman,
* Age > or = 18 years,
* Performance status > or = 1 (according to WHO criteria),
* Patient with histologically proven breast cancer, not metastasized,
* Patient treated with neoadjuvant or adjuvant chemotherapy,
* Absence of cutaneous lesions related to the pathology,
* Patient fluent in the French language,
* Patient affiliated to a social security scheme,
* Obtaining written, signed and dated informed consent.

Exclusion Criteria:

* Metastatic breast cancer,
* Local relapse of breast cancer
* History of cancer in the 5 years preceding the entry into the trial,
* Patient already treated with chemotherapy,
* Medical contraindications to the use of cosmetic products and the prescription of a spa treatment,
* Patient deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Mean satisfaction related to the use of cosmetics during chemotherapy using a visual analog score (VAS) ranging from 0 (not satisfied) to 10 (satisfied). | 6 months
  The mean satisfaction will be assessed using a visual analog score (VAS) ranging from 0 (not satisfied) to 10 (satisfied).
Mean compliance related to the use of cosmetics during chemotherapy by asking if yes or no the products was stopped. | 6 months
  The compliance will be measured by questions asking if patients stopped the use of cosmetics.
Percentage of patients declaring skin problems after the use of these 2 cosmetics | 6 months
  Skin problems will be measured by questions asking if yes or no the skin was moisturized, oily, tugging or nice at touching.
Qualitative assessment of cosmetics : percentage of patients feeling that the products texture/oiliness/application/absorption is good/not good | 6 months
  The qualitative assessment of cosmetics will be measured by questions asking about the texture, the odour, the oiliness, the application and the absorption of the 2 cosmetic products
Patient expectations related to the use of cosmetics during chemotherapy | 6 months
  Patient expectations will be measured by questions asking about the reason why the stopped the use of these 2 cosmetics and by all answers given for the odour, the texture, the oiliness, the application and the absorption

SECONDARY OUTCOMES:
Mean satisfaction related to the use of cosmetics during post-treatment thermal cure using a visual analog score (VAS) ranging from 0 (not satisfied) to 10 (satisfied). | 1 year
  The mean satisfaction will be assessed using a visual analog score (VAS) ranging from 0 (not satisfied) to 10 (satisfied).
Mean compliance related to the use of cosmetics during post-treatment thermal cure by asking if yes or no the products was stopped | 1 year
  The compliance will be measured by questions asking if patients stopped the use of cosmetics
Percentage of patients declaring skin problems after the use of these 2 cosmetics | 1 year
  Skin problems will be measured by questions asking if yes or no the skin was moisturized, oily, tugging or nice at touching.
Qualitative assessment of cosmetics : percentage of patients feeling that the products texture/oiliness/application/absorption is good/not good | 1 year
  The qualitative assessment of cosmetics will be measured by questions asking about the texture, the odour, the oiliness, the application and the absorption of the 2 cosmetic products
Patient expectations related to the use of cosmetics during post-treatment thermal cure | 1 year
  Patient expectations will be measured by questions asking about the reason why the stopped the use of these 2 cosmetics and by all answers given for the odour, the texture, the oiliness, the application and the absorption

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No